CLINICAL TRIAL: NCT01051947
Title: Impact of Nebivolol on Central Aortic Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study already published
Sponsor: Creighton University (Other)
Responsible Party: Jennifer Campbell, PharmD, Creighton University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-15168
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Central Aortic Pressure
Keywords: Nebivolol; Metoprolol; central aortic pressure; hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Experimental): Nebivolol therapy for 2-6 weeks depending on blood pressure readings
  Interventions: Drug: Nebivolol
- Metoprolol (Experimental): Metoprolol therapy for 2-6 weeks depending on blood pressure readings
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Nebivolol — 10 mg by mouth daily for 2 weeks 20 mg by mouth daily for 2 weeks 40 mg by mouth daily for 2 weeks
  Arms: Nebivolol
Drug: Metoprolol — dosage prescribed prior to starting on study
  Arms: Metoprolol

SUMMARY:
A randomized, cross-over, single-blind study to compare the effects of nebivolol and metoprolol on central aortic pressure and peripheral brachial pressure in patients with stable cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with history of hypertension
* Subjects who have received metoprolol for a minimum of 3 months

Exclusion Criteria:

* Patients who have had an acute myocardial infarction, coronary revascularization or who have been hospitalized for heart failure or cardiac arrhythmia in the past 6 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Stable blood pressure | 6 months
  Subjects will be randomized to nebivolol or metoprolol. Their medication will be titrated so that their blood pressure is within 10% of their initial reading.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Campbell, PharmD, Principal Investigator — Creighton University
Locations (1):
- The Cardiac Center at Creighton University, Omaha, Nebraska, United States